CLINICAL TRIAL: NCT02487186
Title: Evaluation of PLGA Microspheres Loaded With Doxycycline Associated to Periodontal Debridement in the Treatment of Chronic Advanced Periodontitis.
Brief Title: Locally Delivered Doxycycline Adjunct to Nonsurgical Periodontal Therapy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Enilson Antonio Sallum, Professor, department of Periodontics, Piracicaba Dental School, State University of Campinas (UNICAMP), Piracicaba, São Paulo, Brazil, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 012/2009
Record Dates: First submitted 2015-06-26; First posted 2015-07-01 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2015-06

CONDITIONS: Periodontal Disease
Keywords: Chronic periodontitis; Local doxycycline; Ultrasonic debridement; PLGA microspheres; Microbiologic assessment
MeSH Terms: conditions — Periodontal Diseases; Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test group: DB+DOX (Active Comparator): Test group: DB (full mouth debridment) +DOX (doxicicline) - 45 minutes of full-mouth debridement + subgingival application of PLGA microspheres loading doxycycline 10%.
  Interventions: Drug: Doxicicline; Procedure: Full-mouth debridment
- Control group: DB alone (Active Comparator): Control group: DB alone (Full-mouth debridment)
  Intervention: 45 minutes of full-mouth debridement + subgingival application of void PLGA microspheres.
  Interventions: Procedure: Full-mouth debridment

INTERVENTIONS:
Drug: Doxicicline — Association of doxycycline (DOX) encapsulated in PLGA microspheres to ultrasonic debridment for the treatment of patients with chronic generalized periodontitis.
  Other Names: PLGA microspheres
  Arms: Test group: DB+DOX
Procedure: Full-mouth debridment — The patients will be treated by a single-session of periodontal debridement
  during 45 minutes, using an ultrasonic instrument (Cavitron, Dentsply, Rio de
  Janeiro, Brazil), under irrigation with sterile saline solution 20. After the debridement, local administration of microspheres loading doxycycline (DOX) (test) or empty microspheres (control) was performed.

SUMMARY:
The aim of this clinical study is to asses the effect of ultrasonic periodontal debridement associated to locally delivered doxycycline (20%) by PLGA microspheres on chronic generalized periodontitis treatment.

DETAILED DESCRIPTION:
Thirty patients with chronic periodontitis and a minimum of seven pockets (>5

mm) in non-molars teeth that bled on probing will be selected. Patients will be randomly

assigned to ultrasonic periodontal debridement followed by local application of doxycycline

by PLGA microspheres (DB+DOX) and periodontal debridement followed by administration

of void PLGA microspheres (DB). Plaque, bleeding on probe, clinical attachment level

(CAL), and probing depth (PD) will be recorded at baseline, 3 and 6 months. Subgingival

biofilm samples will be collected from initially moderate (5 to 6 mm) and deep (≥7 mm)

pockets at baseline, 1, 3 and 6 months. Polimerase chain reaction (PCR) analysis will be

used to detect the frequency of Porphyromonas gingivalis (Pg), Tannerella forsythia (Tf),

Treponema denticola (Td), Aggregatibacter actinomycetemcomitans (Aa), and Prevotella

intermedia (Pi).

ELIGIBILITY:
Inclusion Criteria:

* Chronic generalized periodontitis (AAP,1999);
* At least 7 sites with probing depths >5mm, and 2 sites with probing depth >7mm;
* At least 20 teeth present;
* Systemically healthy.

Exclusion Criteria:

* Had received periodontal care 6 months prior to the study;
* Had taken medications known to interfere with periodontal health and healing 6 months prior to the study;
* Pregnants or lactants;
* Smokers;
* Sensitive to doxycycline.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Probing depht (PD) | 6 months
  Probing depth (PD) will be measured at six sites per tooth by a PCP-15 periodontal Probe (Hu-Friedy - Chicago, IL, USA); This measure will be performed with the use of a plastic stent, presenting edges for the positioning of the stent probe.

SECONDARY OUTCOMES:
Clinical attachment level (CAL) | 6 months
  Six sites per tooth, will be measured with a PCP-15 Periodontal Probe (Hu-Friedy - Chicago, IL, USA). This measure will be performed with the use of a plastic stent, presenting edges for the positioning of the stent probe.

CONTACTS AND LOCATIONS:
Overall Officials: Enilson A Sallum, PhD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Piracicaba Dental School, State University of Campinas, Piracicaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No